CLINICAL TRIAL: NCT01999816
Title: Lifestyle Redesign for Pressure Ulcer Prevention in Spinal Cord Injury
Brief Title: Pressure Ulcer Prevention Study in SCI
Acronym: PUPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Florence Clark, Associate Dean, Chair, and Professor Occupational Science and Occupational Therapy, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-06-00064; R01HD056267 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Spinal Cord Injuries
Keywords: pressure ulcer; lifestyle redesign; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Redesign (Experimental): Occupational therapist led lifestyle redesign program to prevent pressure ulcers
  Interventions: Behavioral: Lifestyle Redesign
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Lifestyle Redesign — Individualized program for lifestyle redesign aimed at decreasing the risk of medically serious pressure ulcers led by licensed occupational therapists trained in the implementation of the lifestyle redesign program
  Other Names: Occupational therapy
  Arms: Lifestyle Redesign

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial of a lifestyle redesign intervention's ability to (1)reduce the incidence of medically serious pressure ulcers and associated surgeries in adults with spinal cord injury, and (2)assess the intervention's cost-effectiveness and potential cost savings and its effects on participants' quality of life.

DETAILED DESCRIPTION:
Medically serious pressure ulcers are a common complication of spinal cord injury (SCI), and are associated with high treatment costs and reduced quality of life. This study will examine the efficacy and cost-effectiveness of a promising lifestyle-based intervention designed to reduce the incidence of pressure ulcers among culturally diverse, community dwelling adults with SCI who have had serious pressure ulcers.

The intervention being tested, termed lifestyle redesign (LR), is based on prior SCI literature as well as on the results of a qualitative pilot study undertaken by our study group. This intervention targets several psychosocial mediating variables that have been shown to be important in prevention of pressure ulcers in daily living contexts. Participants assigned to the LR condition receive individualized in-home sessions, personal phone calls, and incident-based contacts for a 12-month period, followed by 12 months of no intervention. Participants in the control condition do not receive any study-based intervention, but (along with the LR group) have continuing access to the standard options for prevention and treatment that are available through Rancho Los Amigos National Rehabilitation Center.

In addition to identifying a pressure ulcer prevention strategy, the planned research will lead to the development of testable theoretical models of the intervening process mechanisms that link the intervention to pressure ulcer reduction.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (paraplegia or tetraplegia)
* Non-ambulatory
* Able to undergo intervention and testing in English or Spanish
* At least 6 months post-injury
* History of at least one serious (Stage 3 or 4) pressure ulcer in the past 5 years
* Cognitively intact
* Personally expressed willingness to undertake recommended lifestyle changes for ulcer prevention.
* Can be reached by telephone.
* Reside in or within 100 miles of Rancho Los Amigos National Rehabilitation Center (Downey, CA) with no plans to relocate beyond this area.
* Agreement to participate and completion of consent form.

Exclusion Criteria:

* Present serious stage 4 pressure ulcer
* Participation in our preliminary research studies
* Participating in the neuromuscular stimulation study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of serious pressure ulcers | Throughout 12-month study intervention
  New stage 3 or 4 pressure ulcers

SECONDARY OUTCOMES:
Incidence of ulcer related surgeries | Throughout 12-month study intervention and 12-months post intervention period
  Surgical wound repair (flap, skin graft, girdlestone, other)
Quality of life | Throughout 12-month study intervention and 12-months post intervention period
  Measured by the Medical Outcomes Study Short Form (SF-36)
Healthcare service utilization | Throughout 12-month study intervention and 12-months post intervention period
  Estimated cost of healthcare services including inpatient, outpatient, ER, home healthcare, lab, imaging, etc.
Incidence of serious pressure ulcers | Throughout 12-months post intervention period
  New stage 3 or 4 pressure ulcers during the second study year
Life Satisfaction | Throughout 12-month study intervention and 12-months post intervention period
  Measured by the Satisfaction with Life Scale (SWLS)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Clark, PhD, Principal Investigator — University of Southern California; Salah Rubayi, MD, Principal Investigator — Rancho Los Amigos National Rehabilitation Center
Locations (2):
- United States (2):
  - Rancho Los Amigos National Rehabilitation Center (RLANRC), Downey, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified data to ICPSR

REFERENCES:
- [Background] Pyatak EA, Blanche EI, Garber SL, Diaz J, Blanchard J, Florindez L, Clark FA. Conducting intervention research among underserved populations: lessons learned and recommendations for researchers. Arch Phys Med Rehabil. 2013 Jun;94(6):1190-8. doi: 10.1016/j.apmr.2012.12.009. Epub 2012 Dec 21. PMID 23262157
- [Background] Blanche EI, Fogelberg D, Diaz J, Carlson M, Clark F. Manualization of occupational therapy interventions: illustrations from the pressure ulcer prevention research program. Am J Occup Ther. 2011 Nov-Dec;65(6):711-9. doi: 10.5014/ajot.2011.001172. PMID 22214116
- [Background] Vaishampayan A, Clark F, Carlson M, Blanche EI. Preventing pressure ulcers in people with spinal cord injury: targeting risky life circumstances through community-based interventions. Adv Skin Wound Care. 2011 Jun;24(6):275-84; quiz 285-6. doi: 10.1097/01.ASW.0000398663.66530.46. PMID 21586911
- [Background] Fogelberg D, Atkins M, Blanche EI, Carlson M, Clark F. Decisions and Dilemmas in Everyday Life: Daily Use of Wheelchairs by Individuals with Spinal Cord Injury and the Impact on Pressure Ulcer Risk. Top Spinal Cord Inj Rehabil. 2009 Fall;15(2):16-32. doi: 10.1310/sci1502-16. PMID 21603085
- [Background] Clark F, Pyatak EA, Carlson M, Blanche EI, Vigen C, Hay J, Mallinson T, Blanchard J, Unger JB, Garber SL, Diaz J, Florindez LI, Atkins M, Rubayi S, Azen SP; PUPS Study Group. Implementing trials of complex interventions in community settings: the USC-Rancho Los Amigos pressure ulcer prevention study (PUPS). Clin Trials. 2014 Apr;11(2):218-29. doi: 10.1177/1740774514521904. Epub 2014 Feb 26. PMID 24577972
- [Derived] Blanchard J, Vigen C, Mallinson T, Carlson M, Garber SL, Bates-Jensen B. Pressure Injury Data Reconciliation in a Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 Nov;104(11):1833-1839. doi: 10.1016/j.apmr.2023.04.009. Epub 2023 Apr 28. PMID 37121533
- [Derived] Carlson M, Vigen CLP, Rubayi S, Blanche EI, Blanchard J, Atkins M, Bates-Jensen B, Garber SL, Pyatak EA, Diaz J, Florindez LI, Hay JW, Mallinson T, Unger JB, Azen SP, Scott M, Cogan A, Clark F. Lifestyle intervention for adults with spinal cord injury: Results of the USC-RLANRC Pressure Ulcer Prevention Study. J Spinal Cord Med. 2019 Jan;42(1):2-19. doi: 10.1080/10790268.2017.1313931. Epub 2017 Apr 17. PMID 28414254